CLINICAL TRIAL: NCT03719547
Title: Robot-assisted Approach to Cervical Cancer
Acronym: RACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Henrik Falconer, Head of GYN Oncology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS_RACC
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Robot-assisted surgery; Sentinel node biopsy; Laparotomy; Recurrence; Survival
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: Open label, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-assisted radical hysterectomy (Experimental): Total radical hysterectomy with Sentinel lymph node biopsy followed by completion pelvic lymphadenectomy
  Interventions: Procedure: Robot-assisted radical hysterectomy; Diagnostic Test: Sentinel lymph node biopsy
- Abdominal radical hysterectomy (Active Comparator): Total radical hysterectomy with Sentinel lymph node biopsy followed by completion pelvic lymphadenectomy
  Interventions: Procedure: Abdominal radical hysterectomy; Diagnostic Test: Sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Abdominal radical hysterectomy — Radical hysterectomy (type B or C according to the Querleu&Morrow classification) with pelvic lymphadenectomy
  Other Names: TARH; Open radical hysterectomy
  Arms: Abdominal radical hysterectomy
Procedure: Robot-assisted radical hysterectomy — Radical hysterectomy (type B or C according to the Querleu&Morrow classification) with pelvic lymphadenectomy
  Other Names: TRRH; Robotic radical hysterectomy
  Arms: Robot-assisted radical hysterectomy
Diagnostic Test: Sentinel lymph node biopsy — Assessment of sentinel lymph nodes using either radiotracer or indocyanine green (ICG)
  Other Names: SLN

SUMMARY:
The purpose of the RACC trial is to compare the oncologic outcome defined as recurrence-free survival (RFS) between robot-assisted and open radical hysterectomy for the treatment of early stage cervical cancer.

DETAILED DESCRIPTION:
BACKGROUND Cervical cancer is one of the most common female malignancies worldwide, with the largest proportion of women affected in low income countries. Radical hysterectomy with pelvic lymphadenectomy constitutes the primary treatment of early stage cervical cancer. Surgery has traditionally been performed by laparotomy but the past 20 years, the use of minimally invasive techniques has increased. Several studies suggest that laparoscopic radical hysterectomy is associated with less preoperative morbidity and superior quality of life.

In 2005, the Food and Drug Administration (FDA) approved robot-assisted surgery for gynaecological indications. Observational studies have confirmed advantages in form of shorter hospital stay, less bleeding and acceptable OT. Furthermore, compared to conventional laparoscopy OT is significantly shorter with robot technique. Despite wide acceptance and implementation of the robotic system into gynecological oncology todate there are mainly retrospective observational data published on oncological outcomes, offering a low evidence level.

The sentinel node biopsy concept (SNB) is well established in the surgical management of several malignancies including breast, melanoma and vulvar cancer. Theoretically, the implementation would change the management of patients with early cervical cancer dramatically by avoiding multimodal treatment.

Traditionally, radiotracers (Technetium) with or without augmentation of blue dye have been used for SNB. Novel tracers such as fluorescent dyes (indocyanine green (ICG)) have been demonstrated to be superior.

Apart from detection rate, the rate of bilateral mapping of sentinel nodes and sensitivity (false negative rate included), constitutes the most important aspect of the technique. In recent ESGO guidelines on the management of stage IA disease SNB is recommended as the standard treatment unless in patients with positive LVSI where complete PLND should be considered.

RATIONALE In 2018, the LACC (Laparoscopic Approach to Cervical Cancer) trial was completed and the results demonstrated inferiority for minimally invasive surgery (MIS). In the trial, 631 women were randomized to MIS (85% by traditional laparoscopy and the remaining by robot-assisted surgery). Disease-free and overall survival were significantly worse by MIS with no observed advantage in quality of life or perioperative morbidity.

After the trial was closed, two large population-based studies from the Nordic countries (unpublished data) show no difference in either DFS or OS. The absolute majority in these studies were operated by robot-assisted surgery.

Robot-assisted surgery has replaced traditional laparoscopy for radical hysterectomy. Whether robot-assisted surgery is associated with better oncologic outcomes than traditional laparoscopy is unknown.The purpose of the RACC trial is to assess the safety of robot-assisted laparoscopy for the surgical treatment of early stage cervical cancer.

RATIONALE FOR THE QUALITY OF LIFE ASSESSMENT Two randomised controlled trials (LAP2 and LACE) have demonstrated that MIS is superior to laparotomy i in terms of perioperative morbidity and quality of life. However, the LACC trial did not show any differences between MIS and laparotomy for these outcomes. Whether robot-assisted surgery offers superior outcomes is unknown. In the RACC trial, QoL will be assessed in both arms at 5 time points using the EORTC QLQ-CX24 form and the FSFI (Female Sexual Function Index).

RATIONALE FOR THE SENTINEL NODE ALGORITHM Tumor extension to pelvic lymph nodes is the most important prognostic factor in early stage cervical cancer. Traditionally, nodal assessment has been performed through systematic pelvic lymphadenectomy. Sentinel node concepts have been evaluated in several smaller studies but none with sufficient power to properly assess the diagnostic accuracy.

PRIMARY ENDPOINT

- Recurrence-free survival (RFS) at 60 months

SECONDARY ENDPOINTS

* Overall survival (OS) at 60 months
* Perioperative morbidity
* Quality of life
* Diagnostic accuracy of a sentinel node algorithm in cervical cancer
* Health care costs

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma, squamous cell carcinoma or adeno-squamous carcinoma of the uterine cervix;
* Patients with histologically confirmed stage IB (IB3 excluded) and IIA1, according to the latest revision of the FIGO staging manual
* Patients undergoing either a Type B or C radical hysterectomy (Querleu and Morrow classification)
* Patients with adequate bone marrow, renal and hepatic function
* ECOG Performance Status of 0, 1 or 2.
* Patient must be suitable candidates for surgery.
* Patients who have signed an approved Informed Consent
* Age 18 years or older

Exclusion Criteria:

* Any histology other than adenocarcinoma, squamous cell carcinoma or adeno-squamous carcinoma of the uterine cervix
* Tumor size greater than 4 cm
* FIGO stage II-IV (except IIA1)
* Patients with a history of pelvic or abdominal radiotherapy
* Patients who are pregnant
* Patients with contraindications to surgery
* Patients with evidence of metastatic disease by conventional imaging, enlarged pelvic or aortic lymph nodes > 2cm; or histologically positive lymph nodes
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Patients unable to withstand prolonged lithotomy and steep Trendelenburg position
* Patients with secondary invasive neoplasm in the last 5 years (except non-melanoma skin cancer, breast cancer T1N0M0 grade 1 or 2 without any signs of recurrence or activity)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 60 months from surgery
  Time-interval between the date of randomisation and the date of recurrence or the date of death

SECONDARY OUTCOMES:
Overall survival | 60 months from surgery
  Time-interval from the date of randomisation to the date of death (due to any cause), or for patients still alive to the date of last clinical follow-up or contact
Intraoperative complications: number of participants with bowel injuries, urinary tract injuries, hemorrhage requiring vessel suture and/or transfusion, nerve injuries | Complications occurring during intervention (intraoperatively)
  Assessed according to CLASSIC classification and Kaafarani et al.
Post-operative complications: Number of participants requiring pharmacological treatment (CD II) OR surgical, endoscopic or radiological intervention (CD III) OR life-threatening complications requiring ICU-management (CD IV) OR death (CD V) | Postoperative complications are assessed at 30 days postoperatively and at 6 months postoperatively
  Assessed according to the Clavien-Dindo (CD) classification
Health-related quality of life (HRQoL) after surgery for early stage cervical cancer using European Organisation for Research and Treatment of Cancer Quality of Life Cancer Patients (EORTC-QLQ). | Before randomisation, 1 month post surgery, 6 months post surgery, 12 months post surgery, 24 months post surgery, 60 months post surgery
  The response format for the EORTC QLQ is on a four-point scale, from 1 (Not at all) to 4 (Very much). A high score on the functional scales and global quality of life represents a high level of functioning and quality of life. A high score on the symptom scales/items represents a high level of symptoms.
Sentinel lymph node biopsy in cervical cancer | Through study completion, an average of 5 years
  Feasibility of a SLN algorithm: mapping of afferent lymphatic pathways from the cervix to the juxtauterine lymph node. ICG or Technetium99 will be used as tracers.The algorithm comprises removal of suspicious nodes and ultrastaging of sentinel nodes
Health care costs | 6 months from surgery
  Total health care costs including surgical equipment, capital costs, pharmaceuticals, hospitalisation and costs related to re-admission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Falconer, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falconer H, Palsdottir K, Stalberg K, Dahm-Kahler P, Ottander U, Lundin ES, Wijk L, Kimmig R, Jensen PT, Zahl Eriksson AG, Maenpaa J, Persson J, Salehi S. Robot-assisted approach to cervical cancer (RACC): an international multi-center, open-label randomized controlled trial. Int J Gynecol Cancer. 2019 Jul;29(6):1072-1076. doi: 10.1136/ijgc-2019-000558. Epub 2019 Jun 14. PMID 31203203
- See also: Trial website — http://www.racctrial.org